CLINICAL TRIAL: NCT00109057
Title: An Open-Label, Multicenter Extension Study of Recombinant Humanized Monoclonal Anti-VEGF Antibody (rhuMAb VEGF, Bevacizumab) in Subjects Treated With rhuMAb VEGF in a Previous Genentech-Sponsored Phase I or Phase II Cancer Study
Brief Title: An Extension Study to Evaluate Avastin in Patients Treated in a Previous Genentech-Sponsored Cancer Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: AVF0778g
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Cancer
Keywords: Cancer; Advanced malignancies
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab

INTERVENTIONS:
Drug: Avastin (bevacizumab)

SUMMARY:
This is a multicenter, open-label extension study. Subjects who have received rhuMAb VEGF (Avastin) therapy in any Genentech-sponsored Phase I or Phase II cancer study and who did not show evidence of disease progression at completion of the parent study will be eligible for inclusion in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in and completion of a Genentech-sponsored rhuMAb VEGF Phase I or Phase II cancer study
* No evidence of progressive disease at completion of the parent study
* For women of childbearing potential, use of an effective means of contraception
* Signed informed consent

Exclusion Criteria:

* Any unresolved or irreversible rhuMAb VEGF-related ongoing serious adverse events occurring during the parent study
* Any history of central nervous system disease (e.g., primary brain tumor or seizures within 12 months of the first infusion on this study), and/or any evidence of brain metastases
* Compromised renal or hepatic function, as defined in the parent protocol
* Anemia, neutropenia, or thrombocytopenia, as defined in the parent protocol
* Pregnancy (positive pregnancy test) or lactation
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored rhuMAb VEGF cancer study
* Recent (within 3 weeks of the first infusion of this study) major surgical procedure, biopsy of a parenchymal organ, or significant traumatic injury
* Clinically significant cardiovascular disease (e.g., uncontrolled hypertension [blood pressure of >160/110 mmHg on medication], myocardial infarction, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac dysrhythmia requiring medication, or peripheral vascular disease (Grade II or greater)
* Serious, nonhealing wound, ulcer, or bone fracture
* Current or recent (within 10 days of the first infusion on this study) use of oral or parenteral anticoagulants or aspirin (except as required to maintain patency of permanent indwelling intravenous [IV] catheters)
* Inability to comply with study and/or follow-up procedures
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 1998-02; Study Completion 2004-02 (Actual)